CLINICAL TRIAL: NCT05704179
Title: Evaluation of the Relationship Between Obstetric Comorbidity Index and Obstetric Recovery Quality Score in Patients Who Undergo Operative Delivery
Brief Title: Evaluation of the Relationship Between Obstetric Comorbidity Index and Obstetric Quality of Recovery Score
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Gaye Sensoz Celik, Principal investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 23052022162
Record Dates: First submitted 2022-11-14; First posted 2023-01-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life; Obstetric Complication; Cesarean Section Complications; Comorbidities and Coexisting Conditions; Obstetric Anesthesia Problems
Keywords: Obstetric comorbidity index; Obstetric Quality of Recovery; Cesarean section; Obstetric Anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who undergo cesarean section: Obstetric comorbidity index will be calculated for all patients, obstetric quality of recovery score will be evaluated in postpartum period( on the first and second day postpartum)
  Interventions: Other: Obstetric Quality of recovery score

INTERVENTIONS:
Other: Obstetric Quality of recovery score — Patients' quality of recovery will be evaluated with Obstetric Quality of recovery score (ObsQoR-11) on postpartum day 1 and day 2.

SUMMARY:
The goal of this prospective observational study is to learn about the correlation between obstetric comorbidity index and obstetric quality of recovery score in pregnant patients who undergo cesarean section. The main question aims to answer are:

* Are there a correlation between the obstetric comorbidity index and the obstetric quality of recovery score? Can we predict the postoperative quality of recovery by calculating the obstetric comorbidity index before delivery?
* What is the relationship between these scores with the type of anaesthesia given? Participants will answer an 11-question assessment scale to evaluate their recovery of quality in the postpartum period.

DETAILED DESCRIPTION:
After the approval of the ethics committee and the written informed consent of the patients, the patients who are meeting the criteria of inclusion will be included in the study. The demographic data, type of anaesthesia, intraoperative haemorrhage, length of hospital stay and intensive care unit stay(if applicable), the urgency category of the cesarean section, and complications will be recorded. patients will be evaluated with obstetric quality of recovery assessment score on postpartum 1st and 2nd days

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are admitted for Cesarean section > 18 years old
* Speaking Turkish or English
* Agreeing to participate in the study

Exclusion Criteria:

* Pregnant women < 18 years old
* Can not speak Turkish or English
* Not agreeing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Turkish or English-speaking, >18 years old, pregnant patients who undergo cesarean section will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
The correlation between Obstetric comorbidity index (OBCMI) and Obstetric Quality of Recovery score(ObsQoR-11) on postpartum 1st day | each patient will be evaluated on postpartum 1st day
  Obstetric comorbidity index will be calculated before c-section.ObsQoR-11 Questionnaire will be done postoperatively.
The correlation between Obstetric comorbidity index (OBCMI) and Obstetric Quality of Recovery score(ObsQoR-11) on postpartum 2nd day | each patient will be evaluated on postpartum 2nd day
  Obstetric comorbidity index will be calculated before c-section.ObsQoR-11 Questionnaire will be done postoperatively.

SECONDARY OUTCOMES:
Evaluation of the relationship between type of anaesthesia and OBCMI | each patient will be evaluated on the day of c-section
  Type of anaethesia will be recorded from the anaesthesia follow-up sheats. Obstetric comorbidity index will be calculated before c-section.
The relation between Lenght of hospital stay and ObsQoR-11 score on postpartum 1st day | 2months
  Lenght of hospital stay will be recorded from hospital software.ObsQoR-11 will be evaluated on postpartum 1st day
The relation between Lenght of hospital stay and ObsQoR-11 score on postpartum 2nd day | 2months
  Lenght of hospital stay will be recorded from hospital software. ObsQoR-11 will be evaluated on postpartum 2nd day
The relation between complications and OBCMI | 2months
  Complications will be recorded.
The relation between complications and ObsQoR-11 on postpartum 1st day | 2months
  Complications will be recorded
The relation between complications and ObsQoR-11 on postpartum 2nd day | 2months
  Complications will be recorded
The relation between urgency of cesarean section and OBCMI | each patient will be evaluated on the day of c-section
  C-section category will be evaluated
The relation between urgency of cesarean section and ObsQoR-11 score on postpartum 1st day | each patient will be evaluated on the day of c-section
  C-section category will be evaluated
The relation between urgency of cesarean section and ObsQoR-11 score on postpartum 2nd day | each patient will be evaluated on the day of c-section
  C-section category will be evaluated
The relation between intraoperative hemorrhage and OBCMI | On the day of C-section
  Instraoperative hemorrhage will be recorded from the anaesthesia follow-up sheats.
The relation between intraoperative hemorrhage and ObsQoR-11 score on postpartum 1st day | On the day of C-section
  Instraoperative hemorrhage will be recorded from the anaesthesia follow-up sheats.
The relation between intraoperative hemorrhage and ObsQoR-11 score on postpartum 2nd day | The first 2 days postpartum
  Instraoperative hemorrhage will be recorded from the anaesthesia follow-up sheats.
The relation between postoperative intensive care unit stay and OBCMI | each patient will be evaluated on the day of c-section
  Postoperative intensive care unit need and lenght of stay will be recorded
The relation between postoperative intensive care unit stay and ObsQoR-11 score on 1st day | each patient will be evaluated on postpartum 1st day
  Postoperative intensive care unit need and lenght of stay will be recorded.
The relation between postoperative intensive care unit stay and ObsQoR-11 score on 2nd day | each patient will be evaluated on postpartum 2nd day
  Postoperative intensive care unit need and lenght of stay will be recorded.
Demographic data, previous obstetric history and their relation with OBCMI | On the day of C-section
  Demographic data and previous obstetric history will be recorded in preoperative assessment
Demographic data, previous obstetric history and their relation with ObsQoR-11 score on postpartum 1st day | Postpartum 1st day
  Demographic data and previous obstetric history will be recorded in preoperative assessment
Demographic data, previous obstetric history and their relation with ObsQoR-11 score on postpartum 2nd day | Postpartum 2nd day
  Demographic data and previous obstetric history will be recorded in preoperative assessment
Evaluation of the relationship between type of anaesthesia and ObsQoR-11 score on postpartum 1st day | each patient will be evaluated on postpartum 1st day
  Type of anaethesia will be recorded from the anaesthesia follow-up sheats. ObsQoR-11 will be evaluated on postpartum 1st day
Evaluation of the relationship between type of anaesthesia and ObsQoR-11 score on postpartum 2nd day | each patient will be evaluated on postpartum 2nd day
  Type of anaethesia will be recorded from the anaesthesia follow-up sheats. ObsQoR-11 will be evaluated on postpartum 2nd day

CONTACTS AND LOCATIONS:
Overall Officials: Gaye Şensöz Çelik, Principal Investigator — Prof. Dr. Cemil Taşçıoğlu City Hospital
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Result] Bateman BT, Mhyre JM, Hernandez-Diaz S, Huybrechts KF, Fischer MA, Creanga AA, Callaghan WM, Gagne JJ. Development of a comorbidity index for use in obstetric patients. Obstet Gynecol. 2013 Nov;122(5):957-965. doi: 10.1097/AOG.0b013e3182a603bb. PMID 24104771
- [Result] Easter SR, Bateman BT, Sweeney VH, Manganaro K, Lassey SC, Gagne JJ, Robinson JN. A comorbidity-based screening tool to predict severe maternal morbidity at the time of delivery. Am J Obstet Gynecol. 2019 Sep;221(3):271.e1-271.e10. doi: 10.1016/j.ajog.2019.06.025. Epub 2019 Jun 20. PMID 31229427